CLINICAL TRIAL: NCT06865326
Title: Early Detection of Chronic Thromboembolic Pulmonary Hypertension in Patients After Acute Pulmonary Embolism
Brief Title: Early Detection of CTEPH in Patients After APE
Acronym: CTEPH
Status: Recruiting | Type: Observational
Sponsor: Institute of Health Information and Statistics of the Czech Republic (Other Government)
Collaborators: General University Hospital, Prague (Other)
Responsible Party: Sponsor
Other Study IDs: UZIS 2024/2
Record Dates: First submitted 2024-12-02; First posted 2025-03-07 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pulmonary Thromboembolism
Keywords: CTEPH; APE; Early detection; Czech Republic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CTEPH Screening Arm: Patients after APE matching all inclusion & exclusion criteria will undergo a standardized screening process for early detection of CTEPH. The process will include the new screening protocol and in case of a risk of CTEPH, transfer to specialized center for further management.
  Interventions: Other: Standardized CTEPH Screening Protocol

INTERVENTIONS:
Other: Standardized CTEPH Screening Protocol — Implementation of a standardized screening algorithm for early detection of CTEPH in patients after Acute Pulmonary Embolism (APE) and establishment of optimized referral of patients to specialized centers.

SUMMARY:
The project is a national, prospective, multicenter, observational pilot project of screening CTEPH in pacients after APE in the Czech Republic. The main goal of the project is to methodically prepare, implement and evaluate a pilot project that will verify the suitability of the proposed procedure of early detection of Chronic tromboembolic pulmonary hypertesion in such a way as to ensure the maximum positive impact on the health of the population and high cost-effectiveness of the whole process.

DETAILED DESCRIPTION:
The project is a national, prospective, multicenter, observational pilot project of screening CTEPH in pacients after APE in the Czech Republic.

The global goal of the project is to develop, test and implement a uniform procedure for early detection of patients with CTEPH and to set up a process for their rapid referral to a specialized center that treats chronic thromboembolic pulmonary hypertension. The timeliness of the treatment set up has a significant impact on patient's future quality of life and eliminates the risk of subsequent complications or death.

The main objective of this activity is to validate the CTEPH screening process, which will benefit 500 patients in approximately 10 selected centres. Subsequently, patient flow from the cardiologist to a specialised pulmonary hypertension treatment centre will be ensured. The process will include a review and evaluation of the screening algorithm in patients in the pilot.

The project is supported by the European Social Fund (Operational Program Employment plus) and the state budget of the Czech Republic and is registered by the Ministry of Labour and Social Affairs of the Czech Republic under ID: CZ.03.02.02/00/22_005/0002007

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Signed consent to participate in the project and GDPR
* Patients with an episode of acute pulmonary embolism in the last 3-12 months, with ongoing anticoagulation therapy:

  1. Patients with new-onset and ongoing or progressive dyspnea (min. NYHA II) after a pulmonary embolism episode or worsening of dyspnea after a pulmonary embolism episode compared to the status before the episode (at least 1 HYHA grade) or
  2. Asymptomatic patients after a pulmonary embolism episode and at least one of the following risk factors:
* ECHO evidence of severe PH at diagnosis of PE (PASP >60 mmHg)
* Antiphospholipid syndrome with triple positivity (presence of lupus anticoagulans + anti-beta-2-glycoprotein I (B2GPI) antibodies + anticardiolipin)
* Infected permanent venous inlets and cardiac pacing/defibrillation intravascular systems
* Presence of ventriculoatrial shunt for treatment of hydrocephalus
* Nonspecific intestinal inflammation (ulcerative colitis, Crohn's disease)
* History of splenectomy
* Myeloproliferative disorders
* Chronic osteomyelitis

Exclusion Criteria:

* Not agreeing to participate in the project
* Contraindications to treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pacients matching all inclusion & exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Positive predictive value of initial examination | Up to six months from enrollment
  Examinations include echocardiography, CT scan or scintigraphy, and possibly other examinations determined by the cardiologist. Results will be collected from study enrollment to evaluation of all completed examinations by a cardiologist at the primary detection site.
CTEPH detection rates | Up to six months from enrollment
  Results will be collected from study enrollment to evaluation of all completed examinations by a cardiologist at the specialized centre.
Proportion of people with suspected CTEPH who attended a follow-up examination at a specialized pulmonary hypertension treatment centre | Up to six months from enrollment
  Examinations include echocardiography, CT scan or scintigraphy, and possibly other examinations determined by the cardiologist. Results will be collected from study enrollment to evaluation of all completed examinations by a cardiologist at the primary detection site.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Jansa, prof., Study Director — General University Hospital of Prague
Locations (10):
- Czechia (10):
  - Brno University Hospital, Brno
  - Havlíčkův Brod Hospital, Havlíčkův Brod
  - University Hospital Hradec Králové, Hradec Králové
  - Jihlava Hospital, Jihlava
  - Náchod Hospital, Náchod
  - University Hospital Olomouc, Olomouc
  - University Hospital Ostrava, Ostrava
  - Pardubice Hospital, Pardubice
  - Rychnov nad Kněžnou Hospital, Rychnov nad Kněžnou
  - Tábor Hospital, Tábor